CLINICAL TRIAL: NCT01994915
Title: Effects on Functionality of Occupational Therapy Added to Physiotherapy in Severe COPD Patients
Brief Title: Effects of Occupational Therapy in COPD
Acronym: COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, assistant professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF0045UG; FCSDP1010 (Other: Department of Physical Therapy)
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: exacerbation; functionality; occupational therapy; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Occupational Therapy; Activities of Daily Living; Quality of Life

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Occupational therapy group (Experimental): 35 patients diagnosed with chronic obstructive pulmonary disease attending to the Hospital because of an exacerbation are going to be included in this group.
  Interventions: Other: Occupational therapy
- Control group (No Intervention): 35 patients diagnosed with chronic obstructive pulmonary disease are going to be included in this group. They are not going to receive other than standard care (medical and physical therapy intervention).

INTERVENTIONS:
Other: Occupational therapy — Patients included in this group are going to receive an occupational therapy intervention 3 sessions after hospital discharge. The intervention is based on energy conservation techniques improving the execution of the activities of daily living.
  Other Names: Activities of daily living; Functionality; Quality of life; Independence
  Arms: Occupational therapy group

SUMMARY:
Chronic obstructive pulmonary disease is a chronic condition involving an impairment in functionality and in the execution of activities of daily life. The hypothesis of this study is that an occupational therapy intervention added to a physiotherapy program and a medical treatment increase the functionality and the quality of life of patients with chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
The evolution of chronic obstructive pulmonary disease can be aggravated in some periods by an increase of the symptoms (above all, the cough, the dyspnea and the quantity of sputum purulence). This is known as exacerbation, and it is the most frequent reason for hospital stay, urgences services and death in this condition. A physiotherapy program and an occupational therapy intervention are carrying out in patients attending to the Hospital because of an exacerbation.. Participants will be assessed at baseline and again at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic obstructive pulmonary disease with exacerbation.
* No contraindication of physiotherapy.
* Signed written consent.
* Medical approval for inclusion

Exclusion Criteria:

* Heart disease.
* Neurological patients.
* Contraindications of physiotherapy.
* Nursing home residents.
* Cognitive impairments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Functionality | Baseline, 12 months
  Change from baseline to postintervention on functionality. This is assessed using two measures: the Functional Independence Measure and the Canadian Occupational Performance Measure. A follow-up is going to be performed at 1, 3, 6 and 12 months after the occupational therapy intervention.
Quality of life | Baseline, 12months
  Changes from baseline to postintervention in quality of life. It is assessed using two questionnaires, the EuroQoL-5D questionnaire and the Health Questionnaire St. George. A follow-up is going to be performed at 1, 3, 6 and 12 months after treatment.

SECONDARY OUTCOMES:
Anxiety and depression | Baseline, 12 months
  Changes from baseline to postintervention on anxiety and depression measured with the Hospital Anxiety and Depression Scale. Patients are going to complete this questionnaire composed of statements relevant to either generalised anxiety or depression. A follow-up is going to be performed at 1, 3, 6, and 12 months after the intervention.
Activity levels | Baseline, 12 months
  The accelerometer Armband is going to be used for activity monitoring. It measures the intensity of the activity during 12 hours. A follow-up at 1, 3, 6 and 12 months is going to be performed after treatment.
Dyspnoea | baseline, 12 months
  Changes from baseline to postintervention in dyspnoea measured with Borg Scale. A follow-up is going to be performed at 1, 3, 6 and 12 months after occupational therapy treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Department of Physical Therapy, Granada, Spain, Spain